CLINICAL TRIAL: NCT02022150
Title: Body Composition Analysis in Cirrhotic Patients With Ascites Undergoing Paracentesis
Brief Title: Body Composition Analysis in Cirrhotic Undergoing Paracentesis
Acronym: Paracentesis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, ALDO TORRE DELGADILLO, M.D. M.Sc, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Other Study IDs: GAS-819-12/13-1
Record Dates: First submitted 2013-01-17; First posted 2013-12-27 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Liver Cirrhosis; Ascites
Keywords: Paracentesis; Liver Cirrhosis; ascites; body composition
MeSH Terms: conditions — Liver Cirrhosis; Ascites | interventions — Body Composition; Paracentesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Body composition in paracentesis: Taking blood samples and bioelectrical impedance, Psychometric Hepatic Encephalopathy Score (PHES) and Critical Flicker Frequency (CFF) before and after paracentesis.
  Interventions: Behavioral: Body composition in paracentesis

INTERVENTIONS:
Behavioral: Body composition in paracentesis — Takin blood samples and bioelectrical impedance measurmeent, Neuropsychological tests evaluation

SUMMARY:
Ascites is a frequent complication of liver cirrhosis, initial treatment consists on diuretics intake, however, as the disease progresses this complication becomes more severe, consequently other therapeutic options are used.

Paracentesis is indicated when severe ascites is present and it should be accompanied by albumin infusion.

Nutritional status is generally affected in patients with liver cirrhosis, even more patients with severe ascites show decreased energy intake due to gastric compression.

ELIGIBILITY:
Inclusion Criteria:

* Any genre.
* Age 18-70 years old.
* Diagnosis of liver cirrhosis of any etiology (documented by clinical, biochemical, radiological and / or biopsy.
* Presence of high volume ascites
* The signing of informed consent will be required for the inclusion of any patient.

Exclusion Criteria:

* Hepatic encephalopathy grade III or IV. 2) liver transplantation.
* Congestive heart failure.
* Hemodialysis.
* Acute or chronic renal failure.
* Nephrotic syndrome with protein loss.
* Alcoholism active in the last 6 months.
* Pregnancy.
* upper gastrointestinal bleeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The cohort will be selected from the Liver Clinic, Department of Gastroenterology at a tertiary care center in Mexico
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2012-12; Primary Completion 2021-06 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Body composition | Baseline and 8 days post treatment
  bioelectrical impedance vector analysis

CONTACTS AND LOCATIONS:
Overall Officials: Aldo Torre, M.D, M.Sc., Principal Investigator — Instituto Nacional de Nutrición y Ciencias Médicas "Salvador Zubirán"
Locations (2):
- Mexico (2):
  - Instituto Nacional de Ciencias Médicas y Nutrición "Salvador Zubirán", Mexico City, D.F
  - Instituto Nacional de Ciencias Médicas y Nutrición "Salvador Zubirán", Mexico City